CLINICAL TRIAL: NCT05389228
Title: Health Consequences of the Burden of Atrial Fibrillation - The Swiss-AF-BURDEN Study
Brief Title: Health Consequences of the Burden of Atrial Fibrillation
Acronym: SwissAF-BURDEN
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Clinical Trial Unit, University Hospital Basel, Switzerland (Other); Swiss Heart Foundation (Other); Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Michael Kühne, Prof. Dr. med., University Hospital, Basel, Switzerland
Other Study IDs: Swiss-AF-BURDEN
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation; Burden
Keywords: Atrial Fibrillation; Burden
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Swiss-AF-BURDEN study will be embedded in the follow-up visits of the Swiss-AF cohort study. The research question of the current atrial fibrillation burden will be answered by using 7-day Holter-ECG recordings and continuous implanted loop recorder recording, whereas cardiac MRI examination will give results about cardiac dimensions and function. The 7-day Holter ECG will be repeated after one year. The cMRI will be performed separately or directly after the brain MRI to minimize the additional burden for the patients. Only a subsample of 100 patients will additionally receive ILR for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Swiss-AF study patient
* Paroxysmal or persistent AF

Exclusion Criteria:

* Permanent AF
* Swiss-AF patients not willing or able to undergo 7-day Holter monitoring
* Specifically for cMRI: Pregnant women or women of child-bearing age without a prior negative pregnancy test

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from the ongoing Swiss-AF cohort study with paroxysmal or persistent AF
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
AF-burden | Baseline to Follow-up year 2
  The burden of AF is defined as the amount of time (percentage) in AF during rhythm monitoring

SECONDARY OUTCOMES:
Incidence of overt and covert stroke | Baseline to Follow-up year 2
  Number of participants with overt and covert stroke

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kuehne, MD Prof, exec MBA, Principal Investigator — University Hospital, Basel, Switzerland; Laurent Roten, MD Prof, Principal Investigator — University Hospital Insel, Bern, Switzerland; Dipen Shah, MD Prof, Principal Investigator — Hôpitaux Universitaires de Genève, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland